CLINICAL TRIAL: NCT02252861
Title: French Database of Left Atrial Appendage Closure
Acronym: FLAAC
Status: Completed | Type: Observational
Sponsor: Henri Mondor University Hospital (Other)
Collaborators: French association for research in cardiology (ARCARD) (Unknown)
Responsible Party: Principal Investigator, Philippe Le Corvoisier, MD, Henri Mondor University Hospital
Other Study IDs: FLAAC
Record Dates: First submitted 2014-09-22; First posted 2014-09-30 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Atrial Fibrillation and Other Dysrhythmias | Patient
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Left Atrial Appendage Closure: Patients with atrial fibrillation and counter-indication to anticoagulant therapy referred for percutaneous Left Atrial Appendage Closure in routine care
  Interventions: Other: Percutaneous Left Atrial Appendage Closure in routine care

INTERVENTIONS:
Other: Percutaneous Left Atrial Appendage Closure in routine care — The inclusion in the database induces no specific intervention. Percutaneous Left Atrial Appendage Closure is performed for patient care. No specific intervention is performed specifically for the database. Neither left atrial appendage closure procedure nor patient follow up are modified by patient inclusion in the database.

SUMMARY:
Patients with atrial fibrillation are exposed to a high risk of thrombus in the left atrium that can induce cerebral vascular events or systemic embolisms. This justifies the prescription of anticoagulant therapies in patients with high risk of thromboembolic event. Percutaneous left atrial appendage closure is a new interventional strategy for patients with high risk of cardiovascular events and a counter-indication for long term treatment with anticoagulant agents. However, only few data are available on effectiveness and prognosis of patients treated by this new interventional strategy.

This national database record per-procedure and follow-up data of patients treated by left atrial appendage closure.

This database is strictly observational.

Percutaneous left atrial appendage closure is performed only for the purpose of patient care. No specific intervention is performed specifically for the database. Neither left atrial appendage closure procedure nor patient follow up are modified by patient inclusion in the database.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to a french interventional cardiology department for percutaneous left atrial appendage closure in routine care
* Signature of an inform consent form for inclusion of data recorded during care in the database

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred for percutaneous Left Atrial Appendage Closure to one of the French centers involved in this database
Sampling Method: Non-Probability Sample
Enrollment: 840 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Assessment of the rate of thromboembolic events related to atrial fibrillation in patients treated by left atrial appendage closure in daily practice in France | 1 year

SECONDARY OUTCOMES:
Assessment of patient management in daily practice after left atrial appendage closure (number of echocardiography procedures) | 1 year
Death rate from cardiovascular disease after left atrial appendage closure | 1 year
Unexplained Death rate after left atrial appendage closure | 1 year
Adverse events related to the procedure | 1 year
Cost of the procedure of left atrial appendage closure | Costs will be assessed for the duration of hospital stay, an expected average of 3 days
Cost of patient follow-up after left atrial appendage closure | 1 year
Assessment of patient medical treatment in daily practice after left atrial appendage closure (percentage of patients with antiplatelet drugs) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Teiger, MD, PhD, Principal Investigator — emmanuel.teiger@hmn.aphp.fr
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Derived] Teiger E, Thambo JB, Defaye P, Hermida JS, Abbey S, Klug D, Juliard JM, Spaulding C, Armero S, Champagnac D, Bhugaloo H, Ternacle J, Lellouche N, Audureau E, Le Corvoisier P; French national Left Atrial Appendage Closure registry (FLAAC) investigators. Left atrial appendage closure for stroke prevention in atrial fibrillation: Final report from the French left atrial appendage closure registry. Catheter Cardiovasc Interv. 2021 Oct;98(4):788-799. doi: 10.1002/ccd.29795. Epub 2021 May 29. PMID 34051135
- [Derived] Teiger E, Thambo JB, Defaye P, Hermida JS, Abbey S, Klug D, Juliard JM, Pasquie JL, Rioufol G, Lepillier A, Elbaz M, Horvilleur J, Brenot P, Pierre B, Le Corvoisier P; French National Left Atrial Appendage Closure Registry (FLAAC) Investigators. Percutaneous Left Atrial Appendage Closure Is a Reasonable Option for Patients With Atrial Fibrillation at High Risk for Cerebrovascular Events. Circ Cardiovasc Interv. 2018 Mar;11(3):e005841. doi: 10.1161/CIRCINTERVENTIONS.117.005841. PMID 29540492